CLINICAL TRIAL: NCT03066882
Title: Comparison Effects of Negative Calorie Diet and Low-calorie Diet on Weight Loss and Lipid Profile in Sedentary Overweight/Obese Middle-aged and Older Women
Brief Title: Dietary Effects on Weight Loss and Lipid Profile in Sedentary Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: P.L.Shupik National Medical Academy of Post-Graduate Education (Other)
Responsible Party: Principal Investigator, Mohammadreza Rezaeipour, MD, PhD, Assistant professor of sports medicine (sports injury and corrective movement), University of Sistan and Baluchestan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: no grant 3
Record Dates: First submitted 2017-02-17; First posted 2017-03-01 (Actual); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Obesity; Overweight; Life Style
Keywords: Caloric Restriction; Diet; Obesity; Overweight; Sedentary Lifestyle; Weight loss; Women
MeSH Terms: conditions — Obesity; Overweight; Sedentary Behavior; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group I (Experimental): Study group I (19 participants) received the NCD (details of diet: 15% protein, 75% carbohydrates, 10% fat). Both groups had 15% caloric restriction from their maintenance energy requirements.
  Interventions: Dietary Supplement: NCD
- Study group II (Experimental): Study group II (18 participants) received the LCD or healthy weight maintenance diet (details of diet: 15% protein, 55% carbohydrates, 30% fat).Both groups had 15% caloric restriction from their maintenance energy requirements.
  Interventions: Dietary Supplement: LCD

INTERVENTIONS:
Dietary Supplement: NCD — negative calorie diet
  Other Names: group I
  Arms: Study group I
Dietary Supplement: LCD — low calorie diet
  Other Names: group II
  Arms: Study group II

SUMMARY:
Negative-calorie diet is among the popular dieting guides for weight loss; however, there is still little knowledge about this method. The present study aimed to determine the effects of negative-calorie diet on weight loss and lipid profile, and to compare its efficiency with low-calorie diet.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers and weight-stable (± 2 kg, for more than one year) with no history of regular exercise in at least three months before the study.

Exclusion Criteria:

* History of CVD and other disorders such as diabetes, depression, eating disorders, chronic medications, kidney disease, cancer, food allergies or intolerances to items used in meals.
* Subjects with abnormality in thyroid or Electrocardiograph, any history of anti-obesity medication or weight loss drugs or dietary supplementations for weight control.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants were non-smokers and weight-stable (± 2 kg, for more than one year) with no history of regular exercise in at least three months before the study.
Enrollment: 37 (Actual)
Dates: Start 2012-05-10 (Actual); Primary Completion 2015-09-20 (Actual); Study Completion 2016-10-30 (Actual)

PRIMARY OUTCOMES:
Weight | pre-study
  assessed in kg
Total cholesterol (Total-C) | pre-study
  assessed in mg/dl
High-density lipoprotein -cholesterol (HDL-C) | pre-study
  assessed in mg/dl
Low-density lipoprotein -cholesterol (LDL-C) | pre-study
  assessed in mg/dl
Triglycerides (TG) | pre-study
  assessed in mg/dl

SECONDARY OUTCOMES:
Weight | 3-month
  assessed in kg
Total cholesterol (Total-C) | 3-month
  assessed in mg/dl
High-density lipoprotein -cholesterol (HDL-C) | 3-month
  assessed in mg/dl
Low-density lipoprotein -cholesterol (LDL-C) | 3-month
  assessed in mg/dl